CLINICAL TRIAL: NCT03229330
Title: The Effect of Low-level Light Therapy on Treatment of Venous Ulcers Assessed by Nursing Outcomes Classification (NOC): Randomized Clinical Trial
Brief Title: Low-level Light Therapy on Treatment of Venous Ulcers Assesed by Nursing Outcome Classification (NOC)
Acronym: LASERUVe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0634
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2017-07

CONDITIONS: Venous Ulcer; Low-Level Light Therapy
Keywords: Wound Healing; Outcome Assessment (Health Care)
MeSH Terms: conditions — Varicose Ulcer | interventions — Low-Level Light Therapy

STUDY DESIGN:
Masking Description: All subjects involved are aware of the procedures applied due to the features of the therapies used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Low-level Light Therapy: Wavelength of 660 nm (red laser) and Conventional treatment: Topical treatment with compressive therapy, exercises of lower extremities, resting; once a week for 16 weeks.
  Interventions: Procedure: Low-level Light Therapy; Combination Product: Conventional treatment
- Controls (Active Comparator): Conventional treatment: Topical treatment with compressive therapy, exercises of lower extremities, resting; once a week for 16 weeks.
  Interventions: Combination Product: Conventional treatment

INTERVENTIONS:
Procedure: Low-level Light Therapy — Low-level Light Therapy 660nm (red laser), 1 to 3 Joules, irradiation time and number of points varied.
  Other Names: Wavelength of 660 nm; red laser
  Arms: Intervention
Combination Product: Conventional treatment — Topical treatment: essential fatty oil, hydrogel, papain gel, petrolatum gauze, calcium or silver alginate, zinc oxide and barrier cream; and high compression bandage SurePress
  Other Names: Topical and compressive treatments

SUMMARY:
This study compares the effect of adjuvant treatment of Low-level Light Therapy with conventional treatment in the tissue repair of venous ulcers in patients undergoing outpatient nursing consultation. For the evaluation of the cases clinical indicators of Nursing Outcomes Classification have been used.

DETAILED DESCRIPTION:
There are several therapeutics with different mechanisms of action to reach tissue repair.

The conventional treatment of venous ulcers is based on the alternation of exercising the lower extremities with resting, the application of topical treatments associated with compressive therapy, and the use of medications.

Despite the diversity of bandages available, there are still lesions with difficult prolonged healing process. Therefore, Low-level Light Therapy has been used as an adjuvant technological alternative therapy, due to its photochemical effects on the tissues, such as the modulation of inflammation, increase of granulation tissue, contraction of the wound, reduction of the inflammatory process, and reduction of pain. This therapy contributes to accelerate and improve the tissue repair process.

Studies assessed by Nursing Outcomes Classification about the usage of the treatments above combined are not available. Consequently, more robust clinical studies over venous ulcers to evaluate the tissue repair must be proposed using reliable instruments.

ELIGIBILITY:
Inclusion Criteria:

* Presence of venous ulcer
* Availability for weekly appointment
* Acceptance to participate of the research with the signature of the Term of Free and Informed Consent

Exclusion Criteria:

* Morbid obesity
* Active cancer treatment
* Erysipelas
* Cellulitis, lymphangitis and chronic lymphedema
* Usage of immunosuppressants and / or corticosteroids
* Venous ulcer all around the leg
* Presence of coagulation necrosis covering more than 25% of the wound bed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Decreased Wound Size and Scar formation | 16 weeks
  NOC Wound Healing: Second Intention - Greater length (in the cephalopheudial direction) versus greater width, in cm2 evaluated by the Likert scale, being 1 the worst score and 5 best score.
  NOC Wound Healing: Second Intention - Wound covered with epithelial tissue (new pink or bright tissue that develops from the edges or as "islands" on the surface of the lesion) evaluated by the Likert scale, being 1 the worst score and 5 best score.

SECONDARY OUTCOMES:
Skin thickness | 16 weeks
  NOC Tissue Integrity: Skin and Mucous Membranes - Depth reached. It involves layers and structures of the skin altered by loss of tissue integrity (ulcerated area) assessed by the Likert scale, being 1 the worst score and 5 best score.
Evaluation of Pain | 16 weeks
  NOC Tissue Integrity: Skin and Mucous Membranes - Unpleasant sensory and emotional experience arising from actual or potential or described tissue injury, with sudden or slow onset of mild to severe intensity, constant or recurrent, without an anticipated or predictable termination. Evaluated as frequency, condition and intensity by the Likert scale, being 1 the worst score and 5 best score.
Overall improvement of other NOC indicators correlated. | 16 weeks
  Overall improvement of the indicators of NOC results of Wound Healing: Second Intention and Tissue Integrity: Skin and Mucous Membranes.

CONTACTS AND LOCATIONS:
Overall Officials: Amália De Fátima Lucena, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bavaresco T, Pires AUB, Moraes VM, Osmarin VM, Silveira DT, Lucena AF. Low-level laser therapy for treatment of venous ulcers evaluated with the Nursing Outcome Classification: study protocol for a randomized controlled trial. Trials. 2018 Jul 12;19(1):372. doi: 10.1186/s13063-018-2729-x. PMID 30001202